CLINICAL TRIAL: NCT00535431
Title: A Study To Investigate The Effects of AER 001 Administered by Nebulization on Antigen Challenge in Atopic Asthmatic Subjects
Brief Title: Effects of AER 001 Administered by Nebulization on Antigen Challenge in Atopic Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerovance, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QGUY/2005/AER 001/-03; EUDRACT 2005-004829-26
Record Dates: First submitted 2007-09-22; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Allergic Asthma
Keywords: Asthma; allergy; interleukin-4; interleukin-13; IL-4; IL-13
MeSH Terms: conditions — Asthma; Hypersensitivity; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AER 001
  Interventions: Drug: AER 001
- P (Placebo Comparator): sterile saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AER 001 — 60 mg (in nebuliser), twice daily for 28 days
  Other Names: AEROVANT
  Arms: A
Drug: placebo — Sterile saline nebulised, twice daily for 28 days
  Arms: P

SUMMARY:
This is a single centre, double-blind, randomised, parallel group, repeated dose asthmatic subjects. Subjects will receive AER 001 (60 mgs) or placebo twice daily for 28 days. Before and after treatment subjects will be experimentally challenged with inhaled allergen to induce decreases in lung function. The primary outcome is late phase response to allergen as measured by the average percent change in FEV1 from 4-10 hours following allergen. Because AER 001 is a Th2 anti-inflammatory, it is hypothesized that AER 001 treatment will inhibit the late phase response to allergen challenge.

DETAILED DESCRIPTION:
Objectives:

Primary Objective To investigate the effects of AER 001 on the late asthmatic response in mild to moderate asthmatics

Secondary Objectives

* To examine the effects of AER 001 on antigen induced airway hyperactivity to adenosine monophosphate and blood levels of circulating IgE.
* To characterise the pharmacokinetics of nebulised AER 001.

Exploratory Objectives

* To examine the effects of AER 001 on circulating sIL-13Rα2 and IFNgamma.
* To examine the results of single nucleotide polymorphism (SNP) analysis of IL-4, IL-13, IL-4Rα and IL-13R α to determine if there is any correlation between AER 001 response and genotype
* To examine levels of anti-AER 001 following administration of AER 001

Methodology:

* Single centre, double-blind, randomised, parallel group, repeated dose study in male and female asthmatic subjects.
* A sufficient number of subjects (at least 30 subjects) will be recruited to ensure that at least 26 completed sets of data will be obtained.
* Subjects will be randomised to receive either AER 001 60 mg / matched volume Placebo in a ratio of 1 active : 1 placebo ( block size of 6).
* Treatments will be administered by nebulization from a PARI LC Plus nebulizer
* Subjects are to receive b.i.d. administration of AER 001 / placebo for 27 days. A morning dose will be given on Day 28, (24 hours after Day 27 am-dose).

ELIGIBILITY:
Inclusion Criteria:

* • Adult males and females > 18 years.

  * Subjects who if female, are not currently pregnant or breast feeding and are using medically acceptable methods of contraception.
  * Subjects who have a pre study medical history, physical examination, 12 Lead ECG acceptable to the investigator.
  * Subjects who have clinical laboratory tests within the reference ranges or clinically acceptable to the investigator.
  * Subjects who are negative for HbsAg, hepatitis C antibody and HIV II and I test at screening.
  * Subjects who are negative for drugs of abuse and alcohol tests at screening and admission.
  * Positive response on screening to a skin prick test.
  * Adenosine monophosphate PC20 on screening of ≥ 0.04 mg/ml
  * Subjects, who on the Allergen challenge, have a PC20 on allergen and exhibit a late phase response following the allergen challenge.
  * Subjects who have a FEV1 > 70% of predicted.
  * Subjects who have not received steroid treatment in the prior month.
  * Subjects who are non-smokers for at least 3 months prior to screening.
  * Have a < 10 pack year history.
  * Satisfies the Global Initiative in Asthma (GINA, 2002) definition of asthma or have been on treatment for asthma.
  * Subjects with stable, adequately treated medical conditions may be enrolled provided the Principal Investigator does not consider their study participation to place them at increased risk of adverse events. Subjects should continue their concomitant treatments without change during the study.
  * Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

* • Subjects who do not conform to the above inclusion criteria.

  * Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders which would preclude antigen challenge.
  * Subjects who have a clinically relevant surgical history which would preclude antigen challenge.
  * Subjects who have a clinically relevant family history which would preclude antigen challenge.
  * Subjects who have a history of relevant drug hypersensitivity.
  * Subjects who have a history of alcoholism.
  * Subjects who have a history of drug abuse.
  * Subjects who consume more than 28 units (male)/ 21 units (female) of alcohol a week.

(unit = 1 glass of wine = 1 measure of spirits = ½ pint of beer)

* Subjects who have acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn)
* Subjects who have an acute respiratory infection such as influenza at the time of screening and/or admission.
* Female subjects who are not using an acceptable method of contraception.
* Subjects who have used any investigational drug and /or participated in any clinical trial within 3 months of their first dosing.
* Subjects using medication, which in the opinion of the Investigator will affect the outcome of the study.
* Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to first dosing (to review on a case by case basis).
* Subjects who cannot communicate reliably with the investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who have previously taken AER 001

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of AER 001 on the late asthmatic response in mild to moderate asthmatics as measured by average percent fall in FEV1 from 4-10 hours post allergen challenge (i.e. the late phase response)after 28 days of treatment | pre- vs. post 28 days of treatment

SECONDARY OUTCOMES:
Secondary Objectives • To examine the effects of AER 001 on antigen induced airway hyperactivity to adenosine monophosphate and blood levels of circulating IgE. • To characterise the pharmacokinetics of nebulised AER 001. | pre- vs. post 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MD, Principal Investigator — Guy's Drug Research Unit, Quintiles Ltd.
Locations (1):
- Guy's Drug Research Unit, Quintiles, Ltd., London, United Kingdom

REFERENCES:
- [Derived] Slager RE, Hawkins GA, Ampleford EJ, Bowden A, Stevens LE, Morton MT, Tomkinson A, Wenzel SE, Longphre M, Bleecker ER, Meyers DA. IL-4 receptor alpha polymorphisms are predictors of a pharmacogenetic response to a novel IL-4/IL-13 antagonist. J Allergy Clin Immunol. 2010 Oct;126(4):875-8. doi: 10.1016/j.jaci.2010.08.001. No abstract available. PMID 20920778